CLINICAL TRIAL: NCT00563836
Title: Multicenter, Single-arm, Phase II Study of the Trifunctional Antibody Catumaxomab (Anti-EpCAM x Anti-CD3) Administered Intra- and Postoperatively in Patients With Epithelial Ovarian Cancer
Brief Title: Phase II Study of the Trifunctional Antibody Catumaxomab Administered Intra- and Postoperatively in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-CAT-OC-02
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer
Keywords: ovarian cancer; catumaxomab; phase II; intraoperative; adjuvant; trifunctional antibody
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — 10 µg Catumaxomab intraoperatively and 4 ascending doses (10, 20, 50 and 150 µg) on day 7, 10, 13 and 16

SUMMARY:
Primary evaluation of the safety, tolerability and feasibility regarding specific postoperative complications of an adjuvant treatment with catumaxomab administered after tumor resection.

DETAILED DESCRIPTION:
An open label, multi-center, single-arm, phase II study according to Fleming´s one-stage design. The surgical procedure on Day 0 will be performed according to AGO State of the Art, followed by one intraoperative and four postoperative intraperitoneal administrations of catumaxomab within 16 days. The Discharge Visit will be performed when the patient is leaving the hospital but not earlier than 1 day after the last infustion, followed by the End of Study Visit on Day 30.

Catumaxomab is a trifunctional antibody targeting EpCAM on tumor cells and CD3 on T cells. Trifunctional antibodies represent a new concept for targeted anticancer therapy. This new antibody class has the capability to redirect T cells and accessory cells (e.g. macrophages, dendritic cells [DCs] and natural killer [NK] cells) to the tumor site. According to preclinical data, trifunctional antibodies activate these different immune effector cells, which can trigger a complex anti-tumor immune response.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent form before any protocol-specific screening procedures
* patients has a primary diagnosis of an epithelial ovarian cancer including clear cell carcinoma (FIGO IA(G2-G3) - IV)
* Karnofsky index > or equal 70
* female at an age of 18 years or older
* negative pregnancy test

Exclusion Criteria:

* exposure to prior cancer therapy specific for ovarian cancer
* previos treatment with non-humanized mouse or rat monoclonal antibodies
* known / suspected hypersensitivity to catumaxomab or similar antibodies
* second malignangcy within the last 5 years
* presence of constant immunosuppressive therapy
* presence of symptomatic heart failure or occlusive arterial diseases
* inadequate renal or hepatic function
* presence of any acute or chronic systemic infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
the rate of all specific postoperative complications newly observed during a period of 30 days after surgery | 30 days after surgery

SECONDARY OUTCOMES:
safety and efficacy endpoints | EOS is on day 30, post study period additional 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Jahlid Sehouli, MD, Principal Investigator — Klinikum Charité, 13355 Berlin
Locations (2):
- Innsbruck, Austria
- Klinikum Charité, Berlin, Germany

REFERENCES:
- [Background] Burges A, Wimberger P, Kumper C, Gorbounova V, Sommer H, Schmalfeldt B, Pfisterer J, Lichinitser M, Makhson A, Moiseyenko V, Lahr A, Schulze E, Jager M, Strohlein MA, Heiss MM, Gottwald T, Lindhofer H, Kimmig R. Effective relief of malignant ascites in patients with advanced ovarian cancer by a trifunctional anti-EpCAM x anti-CD3 antibody: a phase I/II study. Clin Cancer Res. 2007 Jul 1;13(13):3899-905. doi: 10.1158/1078-0432.CCR-06-2769. PMID 17606723
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051